CLINICAL TRIAL: NCT07308912
Title: Biomodulatory Effects of GaAlAs 940 nm on Pain Control and Wound Healing at Palatal Donor Site Following Free Gingival Graft Harvesting: a Randomized Controlled Clinical Trial
Brief Title: Effect of GaAlAs 940 Laser on Pain and Wound Healing After Free Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Le Thanh Nguyen, Resident Physician, Department of Periodontics, University of Dentistry, HCMC, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1976/ĐHYD-HĐĐĐ
Record Dates: First submitted 2025-12-27; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Low Level Laser Therapy; Healthy; Postoperative Pain Management; Wound Healing
Keywords: low level laser therapy; palatal donor site; free gingival harvesting; pain control; palatal wound healing; photobiomodulation
MeSH Terms: conditions — Agnosia | interventions — Lasers, Semiconductor; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two groups: a laser group receiving adjunctive 940-nm diode laser irradiation in combination with a palatal stent, and a control group receiving a palatal stent alone following free gingival graft harvesting
Who Masked: Outcomes Assessor
Masking Description: Periodontal surgeries are performed by a periodontist with more than 20 years of clinical experience, who is not involved in laser irradiation or clinical outcome assessment. Laser irradiation and digital scanning of the palatal wound area are performed by a trained investigator who does not participate in clinical outcome evaluation. Clinical assessments and measurements of scanned images are conducted by an independent periodontist who is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Laser group (Experimental): After suturing was completed at the recipient site, the donor site in the laser group was irradiated according to the manufacturer's recommended settings. Laser application was performed in the "Pain Therapy" mode using an Epic X diode laser (940 nm wavelength; 0.1 W power; energy density 4 J/cm²; continuous mode; exposure time 40 s; total energy 12 J). The laser beam was held perpendicular to the donor-site wound surface at 0.5 cm, with a spot size of 1 cm². Following irradiation, a palatal stent was placed.
  Interventions: Device: 940 nm GaAlAs diode laser
- Control group (Active Comparator): After suturing was completed at the recipient site. In the control group, only the palatal stent was applied without laser irradiation.
  Interventions: Device: palatal stent

INTERVENTIONS:
Device: 940 nm GaAlAs diode laser — A single session of 940-nm GaAlAs diode laser irradiation is applied to the palatal donor site immediately after free gingival graft harvesting using a continuous, non-contact mode (0.1 W, 4 J/cm² for 40 seconds), in combination with the use of a palatal stent.
  Other Names: Diode laser; Low-level laser therapy (LLLT); Photobiomodulation therapy (PBMT)
  Arms: Laser group
Device: palatal stent — In the control group, only the palatal stent was applied without laser irradiation after suturing was completed at the recipient site
  Arms: Control group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the biomodulatory effects of a 940-nm GaAlAs diode laser on postoperative pain control and wound healing at the palatal donor site following free gingival graft harvesting. Adult patients undergoing free gingival graft surgery will be randomly allocated to receive either a single session of adjunctive diode laser irradiation immediately after surgery or conventional postoperative care alone. Postoperative pain will be assessed using a visual analog scale, while clinical parameters related to wound healing, including bleeding tendency, epithelialization, and wound size reduction, will be evaluated at predefined follow-up time points. The findings of this study may contribute to the clinical understanding of photobiomodulation in free gingival graft surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age;
2. systemically healthy individuals without any conditions that could affect wound healing (e.g., diabetes, immunosuppression, coagulation disorders, Candida infection;
3. full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) <15%;
4. no previous history of palatal tissue harvesting;
5. no use of overdentures or partial dentures covering the donor area.

Exclusion Criteria:

1. pregnant or breastfeeding women;
2. smokers;
3. patients with psychiatric disorders; and
4. patients taking any medications that impair tissue healing and affect pain perception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 2 hours, 3 days, and 7 days after surgery
  Zero is equivalent to no pain and 10 indicates the worst possible pain.
Post-surgical analgesic consumption | Within 3 days after surgery
  The number of 500-mg acetaminophen tablets consumed by participants during the first 3 days after surgery.
Epithelialization of the palatal donor site | Day 7 and 14 after surgery
  Epithelialization at the palatal donor site assessed as a binary outcome (yes/no) using a hydrogen peroxide bubbling test, classified as non-epithelialized (presence of bubbles) or completely epithelialized (absence of bubbles).
Remaining wound area | Immediately after surgery, and 3, 7, and 14 days after surgery
  Changes in palatal donor site wound area measured using serial intraoral digital scans obtained at predefined follow-up time points

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam